CLINICAL TRIAL: NCT00609791
Title: Age-Related Changes in Nanoparticle Albumin Bound (Nab) Paclitaxel Pharmacokinetics and Pharmacodynamics
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients of Different Ages With Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07157; P30CA033572 (NIH); CHNMC-07157; ABRAXIS-ABX206-BC07US; CDR0000586461 (Registry Identifier: NCI PDQ); NCI-2011-02403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)
Record Dates: First submitted 2008-02-06; First posted 2008-02-07 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Taxes; Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel (Experimental)
  Interventions: Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: pharmacological study; Other: physiologic testing; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: cognitive assessment; Procedure: psychosocial assessment and care

INTERVENTIONS:
Drug: paclitaxel albumin-stabilized nanoparticle formulation — 100 mg/m2 3 weeks on 1 week off
Other: pharmacological study — Cycle 1, week 1 at 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 24 and 48 hours
Other: physiologic testing — Prior to treatment, at the end of 2 cycles of therapy and upon completion of therapy
Other: questionnaire administration — Prior to treatment, at the end of 2 cycles of therapy and upon completion of therapy
Other: study of socioeconomic and demographic variables — Prior to treatment, at the end of 2 cycles of therapy and upon completion of therapy
Procedure: cognitive assessment — Prior to treatment, at the end of 2 cycles of therapy and upon completion of therapy
Procedure: psychosocial assessment and care — Prior to treatment, at the end of 2 cycles of therapy and upon completion of therapy

SUMMARY:
RATIONALE: Gathering information from patients of different ages receiving paclitaxel albumin-stabilized nanoparticle formulation for metastatic breast cancer may help doctors understand how the age of the patient changes the way the drug works.

PURPOSE: This phase II trial is studying how well paclitaxel albumin-stabilized nanoparticle formulation works in treating patients of different ages with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine age-related changes in the pharmacokinetics (pK) of weekly paclitaxel albumin-stabilized nanoparticle formulation (nab-paclitaxel) in patients with metastatic breast cancer.
* To determine age-related changes in the pharmacodynamics (toxicity) of nab-paclitaxel in these patients.

Secondary

* To determine response and time to progression in these patients.
* To explore predictors of pK parameters in these patients.
* To explore predictors of the need for dose reduction, dose delays, or grade 3 or 4 toxicity in these patients.

OUTLINE: Patients are stratified by age in years (< 50 vs 50-60 vs 60-70 vs > 70).

Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes once daily on days 1, 8, and 15 as planned. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood is drawn for pharmacokinetic studies periodically during course 1.

Patients complete questionnaires regarding risk factors that would predict for pharmacokinetic parameters at baseline, prior to the third course of treatment, and at end of study. Data collected include medical characteristics, demographics, functional status, comorbidity, psychological status, social functioning and support, nutritional status, and cognition.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of metastatic breast cancer
* Any estrogen receptor, progesterone receptor, or HER-2/neu status allowed as long as the patient will receive paclitaxel albumin-stabilized nanoparticle formulation alone
* First- or second-line chemotherapy treatment for metastatic disease planned

Exclusion criteria:

* Untreated CNS metastases or symptomatic CNS metastases requiring escalating doses of corticosteroids

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (unless bone metastases are present in the absence of liver metastases)
* Bilirubin ≤ 1.5 mg/dL
* Peripheral neuropathy ≤ grade 1
* Creatinine clearance ≥ 30 mL/min (calculated or 24-hour)
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not pregnant or nursing
* No known history of allergic reactions to paclitaxel
* No serious or uncontrolled infection
* Ability to understand and the willingness to sign a written informed consent document

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No ≥ grade 2 toxicity from prior therapy (other than alopecia)
* No taxane for adjuvant therapy or metastatic disease within the past 12 months
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02-11 (Actual); Primary Completion 2011-10-25 (Actual); Study Completion 2026-04-24 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Medical Group, Pasadena, California

REFERENCES:
- [Derived] Hurria A, Blanchard MS, Synold TW, Mortimer J, Chung CT, Luu T, Katheria V, Rotter AJ, Wong C, Choi A, Feng T, Ramani R, Doan CM, Brown J, Somlo G. Age-related changes in nanoparticle albumin-bound paclitaxel pharmacokinetics and pharmacodynamics: influence of chronological versus functional age. Oncologist. 2015 Jan;20(1):37-44. doi: 10.1634/theoncologist.2014-0202. Epub 2014 Dec 9. PMID 25492923

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-paclitaxel
Started | 40
Completed | 39
Not Completed | 1
Not completed — Subject was deemed ineligible after starting study procedures | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 81]
Age, Customized [Count of Participants; unit: Participants]
  <50 | 10
  50-59 | 5
  60-69 | 15
  >=70 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve Over 24 Hours (AUC24)
Description: Mean of area under the curve over 24 hours (AUC24) reported as well as linear regression of AUC24 by age and chemotherapy toxicity risk score.
  Chemotherapy toxicity risk score is based on the following variables and the value assigned to them. Higher scores indicate more risk, range of 2-19:
  patient age (>=72 years); creatinine clearance (<34 mL/min); presence of amenia (<10 g/dL); hearing impairment; falls in the last 6 months; need for assistance with taking medications; limitations in walking one block; decreased social activities; chemotherapy dosing; number of chemotherapy drugs; cancer type
Time Frame: Cycle 1, week 1 at 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours post treatment
Population: Three participants did not have AUC data through 24 hours post treatment due to incomplete blood samples
Measure: Mean (Standard Deviation); unit: µg/mL*hour
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 36
µg/mL*hour | 4711 (2777)
Statistical Analysis 1: Comparison: Nab-paclitaxel; Linear regression of ln AUC24 on age in years; Test type: Superiority; p = 0.055, Regression, Linear; Slope = 0.011, Standard Error of Mean 0.0057
Statistical Analysis 2: Comparison: Nab-paclitaxel; Linear regression of ln AUC24 on chemotherapy toxicity risk score; Test type: Superiority; p = 0.013, Regression, Linear; Slope = 1.17, Standard Error of Mean 0.45

2. Primary Outcome: Mean Clearance (CL)
Description: Mean CL reported as well as regression results of CL by age and chemotherapy toxicity risk score.
  Chemotherapy toxicity risk score is based on the following variables and the value assigned to them. Higher scores indicate more risk, range of 2-19:
  patient age (>=72 years); creatinine clearance (<34 mL/min); presence of amenia (<10 g/dL); hearing impairment; falls in the last 6 months; need for assistance with taking medications; limitations in walking one block; decreased social activities; chemotherapy dosing; number of chemotherapy drugs; cancer type
Time Frame: Cycle 1, week 1 at 0, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 24 hours post treatment
Population: Nine participants did not have CL data due to incomplete blood samples
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 30
L/h | 37.16 (14.81)
Statistical Analysis 1: Comparison: Nab-paclitaxel; Linear regression of ln CL on age in years; Test type: Superiority; p = 0.25, Regression, Linear; Slope = -0.0074, Standard Error of Mean 0.0063
Statistical Analysis 2: Comparison: Nab-paclitaxel; Linear regression of ln CL versus chemotherapy toxicity risk score; Test type: Superiority; p = 0.04, Regression, Linear; Slope = -0.96, Standard Error of Mean 0.44

3. Secondary Outcome: Grade 3 Toxicity Rate by Chemotherapy Toxicity Risk Score
Description: Comparison of presence of grade 3 toxicity rate by risk score distribution.
  Chemotherapy toxicity risk score is based on the following variables. Higher scores indicate more risk, range of 2-19:
  patient age (>=72 years); creatinine clearance (<34 mL/min); presence of amenia (<10 g/dL); hearing impairment; falls in the last 6 months; need for assistance with taking medications; limitations in walking one block; decreased social activities; chemotherapy dosing; number of chemotherapy drugs; cancer type
  Chemotherapy toxicity risk score category:
  Low risk score - toxicity risk score: 0-5 Medium risk score - toxicity risk score: 6-9 High risk score - toxicity risk score: 10-19
Time Frame: Up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
Participants
  Low risk score : Grade 3 toxicity | 5
  Low risk score : No grade 3 toxicity | 25
  Medium risk score : Grade 3 toxicity | 3
  Medium risk score : No grade 3 toxicity | 3
  High risk score : Grade 3 toxicity | 2
  High risk score : No grade 3 toxicity | 1
Statistical Analysis 1: Comparison: Nab-paclitaxel; Test type: Other; p = 0.041, Fisher Exact

4. Secondary Outcome: Best Response
Description: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Assessed after every 2 cycles of therapy until progression, up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
Participants
  Partial Remission | 12
  Stable Disease | 15
  Progressive Disease | 10
  Not evaluable | 2

5. Secondary Outcome: Median Event-free Survival (EFS) in Months
Description: Median and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for EFS. EFS will be estimated using the product limit method of Kaplan and Meier.
  EFS is defined by time to disease recurrence, disease progression or death to due to any cause
Time Frame: From the date treatment begins until the first date on which recurrence, progression or death due to any cause, assessed up to 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
months | 5.7 [3.2 to 9.2]

6. Secondary Outcome: Number of Participants Requiring Dose Reductions
Description: Number of participants requiring a dose reduction is reported and analysis was performed using a student's 2 sample t test to determine the need of dose reductions based on age, AUC, and CL.
Time Frame: At the completion of treatment, up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
Participants | 11
Statistical Analysis 1: Comparison: Nab-paclitaxel; Difference in age based on whether there was need for a dose reduction; Test type: Superiority; p = .38, t-test, 2 sided; Mean Difference (Final Values) = -4.89, 95% CI 2-sided [-16.5 to 6.7]
Statistical Analysis 2: Comparison: Nab-paclitaxel; Difference in AUC24 based on the need of a dose reduction; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.33 to 0.44]
Statistical Analysis 3: Comparison: Nab-paclitaxel; Difference in clearance based on whether there was a need for dose reduction; Test type: Superiority; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = -0.063, 95% CI 2-sided [-0.49 to 0.36]

7. Secondary Outcome: Number of Participants With a Dose Omission
Description: Number of participants with a dose omission is reported and analysis was performed using a student's 2 sample t test to determine the need of dose omission based on age, AUC, and CL.
Time Frame: At the completion of treatment, up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
Participants | 15
Statistical Analysis 1: Comparison: Nab-paclitaxel; Difference in age based on whether there was need for a dose omission; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = 5.81, 95% CI 2-sided [-2.3 to 13.9]
Statistical Analysis 2: Comparison: Nab-paclitaxel; Difference in AUC24 based on whether there was need for a dose omission; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = -0.079, 95% CI 2-sided [-0.39 to 0.23]
Statistical Analysis 3: Comparison: Nab-paclitaxel; Difference in clearance based on whether there was a need for a dose omission; Test type: Superiority; p = 0.51, t-test, 2 sided; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.22 to 0.42]

8. Secondary Outcome: Percent of Participants With a Grade 3 Toxicity
Description: Percent of participants experiencing a grade 3 toxicity is reported and analysis was performed using a student's 2 sample t test to determine the presence of grade 3 toxicity based on age, AUC, and CL.
Time Frame: At the completion of treatment, up to 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nab-paclitaxel
Number analyzed (Participants) | 39
percentage of participants | 26 [13 to 42]
Statistical Analysis 1: Comparison: Nab-paclitaxel; Difference in age based on whether a participant experienced grade 3 toxicity; Test type: Superiority; p = 0.75, t-test, 2 sided; Mean Difference (Final Values) = 1.68, 95% CI 2-sided [-9.3 to 12.7]
Statistical Analysis 2: Comparison: Nab-paclitaxel; Difference in AUC based on whether a participant experienced grade 3 toxicity; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.12 to 0.81]
Statistical Analysis 3: Comparison: Nab-paclitaxel; Difference in clearance based on whether a participant experienced grade 3 toxicity; Test type: Superiority; p = 0.34, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.67 to 0.25]

ADVERSE EVENTS:
Time Frame: Up to 3.5 years
Arm/Group | Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 26/39
Serious Adverse Events (participants affected / at risk) | 2/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel (N=39)
Urinary tract infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-paclitaxel (N=39)
Allergic rhinitis (Immune system disorders) | 4
Hypersensitivity (Immune system disorders) | 1
Immune system disorder (Immune system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hemoglobin decreased (Investigations) | 36
Leukocyte count decreased (Investigations) | 27
Lymphocyte count decreased (Investigations) | 15
Neutrophil count decreased (Investigations) | 19
Platelet count decreased (Investigations) | 7
Atrial fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 8
Edema (General disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 27
Fever (General disorders) | 3
Insomnia (Psychiatric disorders) | 2
Obesity (Metabolism and nutrition disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2
Injection site reaction (General disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash desquamating (Skin and subcutaneous tissue disorders) | 9
Skin disorder (Skin and subcutaneous tissue disorders) | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 3
Hot flashes (Vascular disorders) | 8
Hypothyroidism (Endocrine disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Enteritis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Mucositis (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Typhlitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Hemorrhage (Gastrointestinal disorders) | 3
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Ureteric hemorrhage (Renal and urinary disorders) | 1
Hepatobiliary disease (Hepatobiliary disorders) | 1
Bladder infection (Infections and infestations) | 2
Catheter related infection (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Infectious colitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 1
Small intestine infection (Infections and infestations) | 1
Upper aerodigestive tract infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 4
Infection without neutropenia (Infections and infestations) | 1
Edema limbs (General disorders) | 11
Fibrosis (Musculoskeletal and connective tissue disorders) | 2
Localized edema (General disorders) | 3
Lymphedema (Vascular disorders) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 22
Aspartate aminotransferase increased (Investigations) | 25
Hyperglycemia (Metabolism and nutrition disorders) | 23
Creatine phosphokinase increased (Investigations) | 1
Creatinine increased (Investigations) | 5
Protein urine positive (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hypercholesteremia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 11
Ataxia (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 3
Depressed level of consciousness (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 5
Dizziness (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 19
Tremor (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 5
Eyelid function disorder (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Watering eyes (Eye disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 10
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 11
Breast pain (Reproductive system and breast disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest pain (Cardiac disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Facial pain (General disorders) | 1
Headache (Nervous system disorders) | 7
Joint pain (Musculoskeletal and connective tissue disorders) | 12
Lymph node pain (Blood and lymphatic system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 2
Peritoneal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Urethral pain (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3
Cystitis (Renal and urinary disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Urogenital disorder (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT00609791/Prot_SAP_000.pdf